CLINICAL TRIAL: NCT04044313
Title: Hepatic Arterial Infusion Chemotherapy Plus Lenvatinib and Toripalimab for Advanced Hepatocellular Carcinoma： a Prospective, Single-arm Trial
Brief Title: HAIC Plus Lenvatinib and Toripalimab for Advanced HCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shi Ming (Other)
Responsible Party: Sponsor-Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-S0903
Record Dates: First submitted 2019-08-01; First posted 2019-08-05 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Hepatic artery infusion chemotherapy; Oxaliplatin, 5-Fluorouracil and Leucovorin; Lenvatinib; Toripalimab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC plus Lenvatinib and Toripalimab (Experimental): Hepatic arterial infusion of oxaliplatin , fluorouracil, and leucovorin every 3 weeks. Lenvatinib 12 mg (or 8 mg) once daily (QD) oral dosing. Toripalimab 240mg intravenously every 3 weeks.
  Interventions: Procedure: Hepatic arterial infusion chemotherapy; Drug: Lenvatinib; Drug: Toripalimab

INTERVENTIONS:
Procedure: Hepatic arterial infusion chemotherapy — administration of oxaliplatin , fluorouracil, and leucovorin via the tumor feeding arteries every 3 weeks
Drug: Lenvatinib — 12 mg (or 8 mg) once daily (QD) oral dosing.
Drug: Toripalimab — 240mg intravenously every 3 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of hepatic arterial infusion chemotherapy of oxaliplatin, 5-fluorouracil and leucovorin plus lenvatinib and toripalimab in patients with advanced hepatocellular carcinoma (HCC)

DETAILED DESCRIPTION:
Hepatic arterial infusion chemotherapy (HAIC) of oxaliplatin, 5-fluorouracil and leucovorin was effective and safe for hepatocellular carcinoma. Lenvatinib was non-inferior to sorafenib in overall survival in untreated advanced hepatocellular carcinoma, and programmed cell death protein-1 (PD-1) antibody was effective and tolerable in patients with advanced hepatocellular carcinoma. No study has evaluated HAIC plus lenvatinib and toripalimab. Thus, the investigators carried out this prospective, single-arm study to find out it.

ELIGIBILITY:
Inclusion Criteria:

* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL)
* Patients must have at least one tumor lesion that can be accurately measured according to EASL criteria.
* Barcelona clinic liver cancer-stage C
* Eastern Cooperative Oncology Group performance status of 0 to 2
* With no previous treatment
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Not amendable to surgical resection ,local ablative therapy and any other cured treatment.
* The following laboratory parameters:

Hemoglobin ≥ 8.5 g/dL Total bilirubin ≤ 30mmol/L Serum albumin ≥ 32 g/L ASL and AST ≤ 5 x upper limit of normal Serum creatinine ≤ 1.5 x upper limit of normal INR ≤ 1.5 or PT/APTT within normal limits Absolute neutrophil count (ANC) >1,500/mm3

• Ability to understand the protocol and to agree to and sign a written informed consent document

Exclusion Criteria:

* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of bleeding diathesis.
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known central nervous system tumors including metastatic brain disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Progression free survival rate at 6 months | 6 months
  Progression was defined as progressive disease by independent radiologic review according to RECIST or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS) | 6 months
  OS is the length of time from the date of randomization until death from any cause.
Progression free survival (PFS) | 6 months
  PFS is defined as the time from the date of randomization to the date of the first objectively documented tumor progression or death due to any cause.
Objective response rate (ORR) | 6 months
  ORR, as determined based on tumor response according to RECIST 1.1, is defined as the proportion of all randomized subjects whose best overall response (BOR) is either a CR or PR.
Adverse events | 6 months
  Safety will be evaluated according to the NCI CTCAE Version 4.03. All observations pertinent to the safety of the study medication will be recorded on the CRF and included in the final report.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/35981413